CLINICAL TRIAL: NCT04679779
Title: Effect of Virtual Reality on Selective Motor Control and Upper Limb Functions in Children With Hemiparesis: A Pilot Study
Brief Title: Virtual Reality in Children With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Ebrahem Fayed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: virtual reality
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-01

CONDITIONS: Physical Disability
Keywords: cerebral palsy; selective motor control; upper limb coordination; virtual reality
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Control grouprecivedvDesigned occupational therapy programe including Exercises facilitating hand skill patterns will include basic reach, grasp, carry and release and the more complex skills of in-hand manipulation and bilateral hand use.
  • study group will recieve Wii virtual reality games
  1. Bowling
  2. Frisbee
  3. Basketball
  4. Boxing
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): receive occupational therapy program
  Interventions: Other: designed occupational therapy program
- study group (Experimental): receive wii virtual reality
  Interventions: Other: Wii virtual reality games

INTERVENTIONS:
Other: designed occupational therapy program — Exercises facilitating hand skill patterns will include basic reach, grasp, carry and release and the more complex skills of in-hand manipulation and bilateral hand use.
  Arms: control group
Other: Wii virtual reality games — 1. Bowling
  2. Frisbee
  3. Basketball
  4. Boxing
  Arms: study group

SUMMARY:
children with cerebral palsy have impaired selective motor control and upper limb functions that affect their performance

DETAILED DESCRIPTION:
Twenty volunteer children diagnosed with hemiparetic cerebral palsy will be recruited from national institute of neuromotor system. they will be randomly assigned to intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* - Age between 7 and 11 years
* spasticity grade of 1+ or 2 on MAS
* level I and II on GMFCS
* level II and III on MACS
* Being able to cooperate and being motivated

Exclusion Criteria:

* visual or auditory problems Severe spasticity (an Ashworth spasticity score of 4 in any upper or lower extremities) Severe mental retardation surgeries for spasticity within the past 12 months, toxin injection within the past six months.
* Structural or fixed soft tissue deformities in the affected upper extremity

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Selective voluntary motor control of upper extremity | 6 weeks
  Test of Arm Selective Control will be used to assess selective voluntary motor control of upper extremityIt was developed to quantify the extent to which children with cerebral palsy have selective voluntary motor control. It will be used to assess movement of shoulder, elbow, forearm, wrist, finger and thumb by using simple tools for grasp items from two starting sitting positions

SECONDARY OUTCOMES:
Hand grip strength | 6 weeks
  it will be assessed by hand held dynamometer
- Upper limb function | 6 weeks
  it will be assessed by Bruinink-Oseretsky test for motor proficiency subset 7 of upper limb coordination

CONTACTS AND LOCATIONS:
Overall Officials: hoda eltalawy, professor, Study Chair — Cairo University; shorouk elshennawy, professor, Study Director — Cairo University; amira mahmoud, phd, Study Director — Cairo University
Locations (1):
- Egypt, Giza, Egypt